CLINICAL TRIAL: NCT05052268
Title: A First-in-Human, Multicenter, Phase 1/2, Open-Label Study of XTX202 in Patients With Advanced Solid Tumors
Brief Title: XTX202 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xilio Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XTX202-01/02-001
Record Dates: First submitted 2021-08-23; First posted 2021-09-22 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 XTX202 Dose Escalation and Pharmacodynamics Expansion (Experimental): Part 1A Dose Escalation of XTX202 administered in ascending doses to patients with advanced or metastatic solid tumors to find the recommended phase 2 doses (RP2Ds).
  Part 1B Evaluation of XTX202 in patients with selected advanced solid tumors to further characterize the pharmacodynamic profile of XTX202
  Interventions: Drug: XTX202
- Phase 2 XTX202 Dose Expansion (Experimental): Part 2A will enroll patients with metastatic renal cell carcinoma who have progressed following standard-of-care treatment.
  Part 2B will enroll patients with melanoma who have progressed following standard-of-care treatment.
  Interventions: Drug: XTX202

INTERVENTIONS:
Drug: XTX202 — XTX202 Monotherapy

SUMMARY:
A First-in-Human, Multicenter, Phase 1/2, Open-Label Study of XTX202 in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/2, multicenter, open-label study designed to evaluate the safety, tolerability, and efficacy of XTX202, an engineered IL-2 prodrug with its activity masked, as monotherapy in patients with advanced solid tumors.

Phase 1 Part 1a will examine XTX202 monotherapy in an accelerated and standard 3+3 dose-escalation design. Based on the results of Part 1a, Part 1b will be initiated to further examine XTX202 in patients with select advanced solid tumors and to further characterize XTX202.

Based on results of Phase 1 patients with select advanced solid tumors will be enrolled in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Disease Criteria

   * Phase 1, Part 1a: Any histologically or cytologically confirmed solid tumor malignancy that is locally advanced or metastatic and has failed standard therapy, or standard therapy is not curative or available
   * Phase 1, Part 1b: Histologically or cytologically confirmed solid tumor malignancy with one of the following tumor histologies: RCC of clear cell histology only, melanoma, squamous cell skin carcinoma, ovarian cancer, non-small cell lung cancer. Those patients who previously received immunotherapy must have derived benefit from this treatment. Additionally, patients with any of the above histologies in an advanced setting who plan to undergo debulking surgery or oligometastasectomy may be eligible to receive 2 cycles of XTX202 treatment in a "window of opportunity" subcohort".
   * Phase 2, Part 2a: Patients with metastatic RCC who have previously been treated with an anti-PD-1 and a TKI, per local and institutional SOC. Patients must have progressed on treatment with an anti-PD-1 mAb administered either as monotherapy or in combination with other therapies
   * Phase 2, Part 2b: Patients with unresectable or metastatic melanoma who have previously been treated with at least 1 prior line of therapy in the recurrent or metastatic setting. Prior therapy must have included an anti-PD-1 alone or in combination per local and institutional standard of care, and patient must have progressed on checkpoint inhibitor therapy. Patients with BRAF V600-activating mutation must have previously received targeted therapy per local and institutional standard of care.
2. ECOG performance status of 0 or 1
3. Adequate organ function
4. Part 1b only patients must be willing to provide fresh tumor biopsies before and after initiation of study treatment.

Exclusion Criteria:

1. Received prior treatment with IL-2 therapy
2. History of clinically significant pulmonary disease
3. History of clinically significant cardiovascular disease
4. Has a diagnosis of immunodeficiency
5. Has an active autoimmune disease that has required systemic treatment in past 2 years, including the use of disease modifying agents, corticosteroids or immunosuppressive drugs
6. Has an active infection requiring systemic therapy within 4 weeks prior to study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) (Phase 1 Part 1A only) | Cycle 1 day 1 up to just prior to the second dose of study drug at Cycle 2 day 1 (each cycle is 21 days)
Incidence of treatment-emergent adverse events (Phase 1 only) | Up to 24 months
Incidence of changes in clinical laboratory values (Phase 1 only) | Up to 24 months
Investigator-assessed objective response rate (ORR) per RECIST 1.1 (Phase 2 only) | Up to 24 months

SECONDARY OUTCOMES:
Plasma concentrations of XTX202 (total and intact) | Up to Cycle 7 (21 days per cycle)
Maximum observed plasma concentration (Cmax) | Up to Cycle 7 (21 days per cycle)
Time of maximum observed concentration (Tmax) | Up to Cycle 7 (21 days per cycle)
Trough concentrations (Ctrough) | Up to Cycle 7 (21 days per cycle)
Area under the curve (AUC) | Up to Cycle 7 (21 days per cycle)
Half-life (T1/2) | Up to Cycle 7 (21 days per cycle)
Systemic clearance (CL) | Up to Cycle 7 (21 days per cycle)
Volume of distribution (Vd) | Up to Cycle 7 (21 days per cycle)
Antidrug antibody (ADA) occurrence and titer in serum (Phase 1 only) | Up to 24 months
Investigator-assessed objective response rate (ORR) per RECIST 1.1 (Phase 1 only) | Up to 24 months
Duration of response (DOR) (Phase 2 only) | Up to 24 months
Disease control rate (Phase 2 only) | Up to 24 months
Progression-free survival (PFS) (Phase 2 only) | Up to 24 months
Overall survival (OS) (Phase 2 only) | Up to 24 months
Incidence of treatment-emergent adverse events (Phase 2 only) | Up to 24 months
Incidence of changes in clinical laboratory values (Phase 2 only) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian- Newport Beach, Newport Beach, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - HealthPartners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - The Ohio State University Wexner Medical Center James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - UPMC Hillman Cancer Center Pavilion, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No